CLINICAL TRIAL: NCT00054314
Title: An Uncontrolled, Phase II Study Evaluating Anti-Tumor Efficacy and Safety of BAY 59-8862 in Patients With Taxane Resistant Non-Small Cell Lung Carcinoma (NSCLC)
Brief Title: BAY 59-8862 in Treating Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Masking: None | Purpose: Treatment
Other Study IDs: DS 02-04; RPCI-DS-0204; BAYER-10653
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — IDN 5109

INTERVENTIONS:
Drug: ortataxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of BAY 59-8862 in treating patients who have non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall response rate, including partial and complete response, in patients with taxane-resistant non-small cell lung cancer treated with BAY 59-8862.
* Determine the overall survival of patients treated with this drug.
* Determine duration of response and time to progression in patients treated with this drug.
* Determine the quantitative and qualitative toxic effects of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive BAY 59-8862 IV over 1 hour on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients with responding disease receive 2-4 additional courses beyond maximal response.

Patients are followed every 3 months for 2 years and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 14-84 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer
* Measurable disease

  * A CNS lesion cannot be the sole target lesion
* Must be taxane-resistant as defined by the following criteria:

  * At least 1 prior course (3 weeks of continuous therapy) of a taxane
  * Progressive disease developed either during or within 6 months after therapy
* No metastatic brain or meningeal tumors unless the following criteria apply:

  * More than 6 months since definitive therapy
  * Negative imaging study within the past 4 weeks
  * Clinically stable with respect to the tumor
  * No concurrent acute steroid therapy or taper

    * Chronic steroids allowed provided dose is stable for 1 month before and after screening radiography

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT and AST no greater than 2.5 times ULN (5 times ULN if liver involvement)
* No chronic hepatitis B or C

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* No congestive heart failure
* No serious cardiac arrhythmias
* No active coronary disease or ischemia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* HIV negative
* No active clinically serious infection
* No history of seizure disorder

  * History of seizures related to brain metastasis allowed if seizure free for the past 2 months
* No prior hypersensitivity to taxane compounds that was unmanageable with premedication
* No pre-existing peripheral neuropathy greater than grade 1
* No other malignancy within the past 3 years except carcinoma in situ of the cervix, adequately treated basal cell carcinoma, or superficial bladder tumors (Ta, Tis, and T1)
* No substance abuse
* No medical, psychological, or social condition that would preclude study participation or evaluation
* No condition that is unstable or would jeopardize patient safety and study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 3 weeks since prior anticancer immunotherapy
* More than 3 weeks since prior biologic response modifiers (e.g., filgrastim [G-CSF])
* More than 4 months since prior bone marrow transplantation or stem cell rescue
* No concurrent anticancer immunotherapy
* Concurrent epoetin alfa allowed if dose is stable for the past 2 months

Chemotherapy

* See Disease Characteristics
* More than 3 weeks since prior anticancer chemotherapy (6 weeks for mitomycin or nitrosoureas)
* No more than 2 prior anticancer chemotherapy regimens (adjuvant therapy is not included unless cancer recurred during or within 6 months after completion of adjuvant therapy)
* No prior oxaliplatin
* No other concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* More than 3 weeks since prior radiotherapy
* No concurrent non-palliative radiotherapy

  * Palliative radiotherapy allowed provided that all of the following criteria are met:

    * No progressive disease
    * No more than 10% of the bone marrow is irradiated
    * Radiation field does not encompass a target lesion

Surgery

* More than 4 weeks since prior surgery
* No prior organ allograft

Other

* More than 4 weeks since prior investigational drug therapy
* No concurrent non-conventional therapies (e.g., herbs or acupuncture) or vitamin/mineral supplements that would interfere with study endpoints
* No other concurrent investigational drug therapy
* No other concurrent anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-03; Primary Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nithya Ramnath, MD, Study Chair — Roswell Park Cancer Institute